CLINICAL TRIAL: NCT07094880
Title: Study on the Use of Subcuteous Use of Methotrexate in Patients With Active Rheumatoid Arthritis
Brief Title: Subcuteous Methotrexate in Rheumatoid Arthritis
Acronym: SCMTXRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangladesh Medical University (Other)
Responsible Party: Principal Investigator, Dr Md. Masudul Hassan, Associated Professor, Bangladesh Medical University, Bangladesh Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 712/2013
Record Dates: First submitted 2025-05-29; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Methotrexate Adverse Reaction; Advantage of Using Subcutaneous Route for Methotrexate
Keywords: Oral Methotrexate; Subcutaneous Methotrexate; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Oral Methotrexate 25 mg will be given weekly
  Interventions: Drug: Tab. Methotrexate 25mg/week
- Group B (Active Comparator): Subcutaneous methotrexate will be given 25mg/week
  Interventions: Drug: Inj. Methotrexate 25mg/week

INTERVENTIONS:
Drug: Tab. Methotrexate 25mg/week — Tab. Methotrexate will be given orally in one arm at a dose of 25 mg/week
  Arms: Group A
Drug: Inj. Methotrexate 25mg/week — Inj. Methotrexate 25 mg/week will be given subcutaneously in another arm
  Arms: Group B

SUMMARY:
Methotrexate use is important for the treatment of Rheumatoid arthritis. Some patients can not tolerate oral methotrexate. So subcutaneous may help to overcome it.

DETAILED DESCRIPTION:
Objective: To see the efficacy and safety of subcutaneous (SC) methotrexate (MTX) in patients suffering from active rheumatoid arthritis (RA). Methods: This was an open labeled randomized clinical trial. Total 90 patients were enrolled from out-patient and in-patients department of medicine (Rheumatology wing) Bangabandhu Sheikh Mujib Medical University. This study was done in two phases. In phase 1, after enrollment 10 mg MTX was given to all patients. After 4 weeks, the dose of MTX was increased by 5 mg. All patients were followed up at 8 weeks from enrollment for outcome measures and tolerability. In phase 2, patients who are intolerant to oral MTX will received 20 mg MTX subcutaneously (n=40). After 8 weeks the dose of MTX was increased by 5 mg. So, 25 mg MTX was given and after another 8 weeks final follow up was given both for clinical and laboratory outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patient must fulfill the ACR 1987 revised criteria
* The disease should be active
* Age 18-70 years

Exclusion Criteria:

* Presence of other rheumatologic disorder
* Pregnancy, lactating mother and women with child bearing potential failing to confirm adequate contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology 20 | "From enrollment to the end of treatment at 16 weeks"
  20% reduction in disease activity

IPD SHARING:
Plan to Share IPD: Undecided